CLINICAL TRIAL: NCT05759819
Title: An Exploratory Study to Evaluate the Efficacy and Safety of the Cilostazol-coated BioMimics 3D Stent System in Patients with Peripheral Occlusive Arterial Disease
Brief Title: Evaluate the Efficacy and Safety of the Cilostazol-coated BioMimics 3D Stent System in Patients with Peripheral Arterial Occlusive Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Otsuka Medical Devices Co., Ltd. Japan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVT-22-001
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CLZ-BM3D group (Experimental): The cilostazol-coated BioMimics 3D stent on the delivery system is implanted into the target lesion and self-expands to maintain the vessel lumen diameter. Post-dilatation is performed as needed.
  - CLZ is released from the surface of the implanted stent.
  Interventions: Device: Standard stenting

INTERVENTIONS:
Device: Standard stenting — The cilostazol-coated BioMimics 3D stent on the delivery system is deployed into the target lesion.

SUMMARY:
An exploratory evaluation of the efficacy and safety of CLZ-BM3D for the treatment of symptomatic peripheral occlusive arterial disease of the superficial femoral artery or proximal popliteal artery

DETAILED DESCRIPTION:
This Study demonstrate an exploratory evaluation of the efficacy and safety of CLZ-BM3D for the treatment of symptomatic peripheral occlusive arterial disease of the superficial femoral artery or proximal popliteal artery

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ankle-brachial index (ABI) of 0.90 or less in the target lower extremity at rest.
* Patients with stenotic lesions (target lesions) requiring treatment of SFA or PPA.
* Patients with Rutherford classification 2, 3, or 4.
* The reference vessel diameter of the target lesion is between 4 mm or more and 5 mm by operator's visual estimate.
* The total length of target lesion measure ≦50㎜ by operator's visual estimate.
* Target lesion lumen stenosis is >70% diameter stenosis by operator's visual estimate.

Exclusion Criteria:

* Patients with a history of surgical or endovascular treatment (including any percutaneous transluminal balloon angioplasty, stenting, atherectomy, or bypass) of the target lesion or vessel prior to enrollment in this study.

However, a history of balloon dilatoplasty with POBA is acceptable if it was performed earlier than 12 months prior to enrollment.

* Patients with a history of major amputation of the target lower extremity.
* Patients with another stenotic lesion in the target or contralateral lower extremity other than the target lesion that is judged to require surgery or endovascular treatment at the time of consent or within 12 months after the procedure.

However, if the patient has another stenotic lesion in the iliac artery other than the target lesion, treatment of the iliac artery lesion (POBA and stenting) is allowed at the time of the study procedure.

* Patients with acute coronary syndrome or stroke/cerebrovascular event within 3 months prior to obtaining consent.
* Patients with coagulopathy.
* Patients with renal insufficiencyor on dialysis.
* Patient who administered orally cilostazol within 7 days prior to the study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary patency of stent at 12 months after the investigational procedure | 12 months
  Loss of primary patency of the stent is determined as any of the following cases.
  * The case as the peak systolic velocity ratio (PSVR) exceeds 2.4
  * The case as the subject had a CDTLR.
  * The case as the angiography revealed > 50% lumen diameter stenosis.
Composite of major adverse events (MAEs) up to 12 months after the investigational procedure | 12 months
  MAE is defined as :
  * All death within 30 days after the study procedure.
  * Major amputation of target lower extrimity
  * Clinically driven target lesion revascurarization.

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu, Chiba
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Osaka Keisatsu Hospital, Osaka City, Osaka

IPD SHARING:
Plan to Share IPD: No